CLINICAL TRIAL: NCT04696757
Title: Non-OpeRative MANagement of Rectal Cancer Patients Who Had Clinical Complete Response After Pre-operative Chemo-raDiotherapY
Brief Title: Non-OpeRative MANagement of Rectal Cancer Patients
Acronym: NORMANDY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Dong-Hoe Koo, Professor, Kangbuk Samsung Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NORMANDY
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Rectal Cancer; Chemoradiotherapy; Watch & Wait
Keywords: Rectal Cancer; Chemoradiotherapy; Watch & wait; Capecitabine
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Intervention Model Description: Aim: 1) to analyze the treatment results after receiving capecitabine adjuvant chemotherapy for 4 months after non-surgical treatment in patients who had completed and could have clinical complete remission with capecitabine preoperative chemoradiotherapy with capecitabine for mid-to-lower rectal cancer 2) to investigate the feasibility of non-surgical treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cape (Experimental): Capecitabine without surgery
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — Capecitabine without surgery

SUMMARY:
This study is a single-center, open, prospective, single-treatment trial (pilot study). This study aims to analyze the treatment results after receiving capecitabine adjuvant chemotherapy for 4 months after non-surgical treatment in patients who had completed and could have clinical complete remission with capecitabine preoperative chemoradiotherapy with capecitabine for mid-to-lower rectal cancer and to investigate the feasibility of non-surgical treatment.

DETAILED DESCRIPTION:
Indication:

1. mid-to-lower rectal cancer was diagnosed histologically as adenocarcinoma in preoperative examination,
2. the tumor was located at the lower boundary of the tumor spans the anorectal junction, and the clinical stage is stage 2 or 3, and
3. clinical complete remission was confirmed after the treatment response evaluation at 8 weeks after completion of preoperative chemoradiotherapy according to MR/SFS and biopsy.

Aim:

1. to analyze the treatment results after receiving capecitabine adjuvant chemotherapy for 4 months after non-surgical treatment in patients who had completed and could have clinical complete remission with capecitabine preoperative chemoradiotherapy with capecitabine for mid-to-lower rectal cancer
2. to investigate the feasibility of non-surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical CR after pre-operative CRT for Rectal cancer

Exclusion Criteria:

-

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
DFS | Duration from Pre-operative CRT
  Disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Hoe Koo, Principal Investigator — Kangbuk Samsung Hospital, Sungkyunkwan University School of Medicine
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No